CLINICAL TRIAL: NCT04348565
Title: An Evaluation of the Effect of a Diabetes Care Programme for People With Type 2 Diabetes Mellitus in Primary Care Setting: A Randomized Controlled Trial
Brief Title: Diabetes Care Programme for Type 2 Diabetes Mellitus in Primary Care Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Association of Hong Kong Nursing Staff (Unknown)
Responsible Party: Principal Investigator, Hau Yee CHUNG, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CREC2019.290; Clinical Research Ethics (Other: Joint CUHK-NTEC CREC)
Record Dates: First submitted 2020-04-05; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Care Programme; Diabetes Conversation Map; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Care Provider
Masking Description: single-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes Care Programme (Experimental): People with Type 2 Diabetes Mellitus of private general practitioner (GP) with solo-practice who receive the intervention (Diabetes Care Programme) in addition to usual medical care at the GP
  Interventions: Other: Diabetes Care Programme
- Standard Usual Care (No Intervention): People with Type 2 Diabetes Mellitus of private general practitioner (GP) with solo-practice who only receive the usual medical care at the GP

INTERVENTIONS:
Other: Diabetes Care Programme — 20-week Diabetes Care Programme consists of three Diabetes Conversation Map sessions in 8 weeks with 3-4 weeks intervals, then two teleconsultations at week 12th and week 16th
  Arms: Diabetes Care Programme

SUMMARY:
Uncontrolled metabolic parameters and co-morbidity risk factors cause Diabetes Mellitus as the leading cause of a multitude of micro-/macro-vascular complications. According to the International Guidelines and Recommendations, people with Type 2 Diabetes Mellitus (T2DM) should attend diabetes educational programmes periodically and optimize the metabolic index of control. In Hong Kong, General Practitioners with solo-practice (GP-SP) have the least availability of resources and support in DM management. A discrepancy of diabetes care between public and private settings and a gap of clinical practice between public-private healthcare settings is identified. In relation to the big population of T2DM is caring by GP-SP but no structured Diabetes Care Programme (DCP) is in place. A structured DCP for T2DM is in need to fill up the clinical gap and make beneficial to the target subjects.

The aim of this study is to evaluate the effectiveness of a DCP for people with T2DM in primary care settings. It is a multi-center, single-blind randomized controlled trial with parallel groups pre-test and post-test design. The evidence-based intervention (DCP) will be carried out in a private primary care setting. People with T2DM attending the GP-SP who meet the study criteria will be randomly assigned into one of the two study groups, either "DCP in addition to usual medical care" or "Usual medical care only" as a control group. The intervention group can beneficial in clinical and psychosocial outcomes after the completion of the 20-week structured DCP with a greater improvement of HbA1c level, Self-Efficacy in diabetes management, Diabetes Empowerment level, Diabetes Knowledge, and Quality of Life than those who only received usual medical care at the GP-SP.

DETAILED DESCRIPTION:
This study is to implement an evidence-based develop Diabetes Care Programme (DCP) for 152 adults with Type 2 Diabetes Mellitus (T2DM) in a few clinics of a general practitioner with solo-practice (GP-SP) in community, and evaluate its effectiveness by comparing the outcomes between study group (DCP with the usual medical care) and control group (Usual medical care only). It is believed that a structured DCP can promote greater clinical outcomes improvement and behavioral changes in the study group as evidence showed in literature. The primary outcomes are glycemic control (HbA1c level) and Self-Efficacy in diabetes management; whereas Diabetes Empowerment level, Diabetes Knowledge and Quality of Life are the secondary outcomes.

The DCP consists of two parts, conduct 3 interactive group education with an innovative educational tool "Diabetes Conversation Map™" sessions by dietitian and diabetes educator/nurse. Then it followed by another 8 weeks for delivering two 15-30 minutes teleconsultations for patient empowerment and follow-up of "Action Plan" by a diabetes educator/nurse. Evaluation of outcomes will be done before the DCP (baseline), at week-8 (right after the group sessions), and at week-20 (4 weeks after the last teleconsultation).

In addition, a focus group interview will be carried out after the completion of the whole intervention. It purposes to explore and get valuable descriptive information and feelings from participants about the intervention and diabetes self-management.

ELIGIBILITY:
Inclusion Criteria:

1. People with T2DM and follow up at private general practitioner
2. Age 18-75
3. Haemoglobin A1c (HbA1c) >7.0%
4. Can communicate in Cantonese

Exclusion Criteria:

1. Insulin users
2. Unstable emotional and/or mental status
3. Cognitive impairment and/or learning disabilities
4. Recruited in other research and/or diabetes educational programme during the study period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Glycated haemoglobin (HbA1c) | Change from Baseline HbA1c at week 20
  Glycemic control
Self-efficacy level in diabetes management | Change from Baseline Self-efficacy level at week 8
  To assess the Self-efficacy level in diabetes management of Chinese people with diabetes. Includes 20 items of self-care in six domains with 1-10 rating scale. Higher score means better self-care.
Self-efficacy level in diabetes management | Change from Baseline Self-efficacy level at week 20
  To assess the Self-efficacy level in diabetes management of Chinese people with diabetes. Includes 20 items of self-care in six domains with 1-10 rating scale. Higher score means better self-care.

SECONDARY OUTCOMES:
Diabetes Empowerment Scale | Change from Baseline Psycho-social Self-efficacy level at week 8
  To assess the overall psycho-social self-efficacy level of Chinese people with diabetes. It includes 10 items with a 1-5 rating scale. A higher score means a higher level of self-efficacy.
Diabetes Empowerment Scale | Change from Baseline Psycho-social Self-efficacy level at week 20
  To assess the overall psycho-social self-efficacy level of Chinese people with diabetes. It includes 10 items with a 1-5 rating scale. A higher score means a higher level of self-efficacy.
Diabetes Knowledge Questionnaire | Change from Baseline Diabetes self-care knowledge at week 8
  To assess the Diabetes self-care knowledge of Chinese people with diabetes. It includes 24 items of diabetes self-care knowledge with the total score range from 0-24. Valid responses with "yes", "no" or "I don't know"; only scored on correct answers. A higher score means a higher level of diabetes knowledge.
Diabetes Knowledge Questionnaire | Change from Baseline Diabetes self-care knowledge at week 20
  To assess the Diabetes self-care knowledge of Chinese people with diabetes. It includes 24 items of diabetes self-care knowledge with the total score range from 0-24. Valid responses with "yes", "no" or "I don't know"; only scored on correct answers. A higher score means a higher level of diabetes knowledge.
Quality of life Measurement | Change from Baseline Quality of Life status at week 8
  The valuation of health status (quality of life) of Chinese people. It includes 5 health dimensions with a sum of negative validity & 1 visual analog scale to reflect the self-rated health score. A higher score means a higher quality of life status.
Quality of life Measurement | Change from Baseline Quality of Life status at week 20
  The valuation of health status (quality of life) of Chinese people. It includes 5 health dimensions with a sum of negative validity & 1 visual analog scale to reflect the self-rated health score. A higher score means a higher quality of life status.

CONTACTS AND LOCATIONS:
Overall Officials: Hau Yee H CHUNG, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Clinics of private general practitioners, Hong Kong, Hong Kong SAR, Hong Kong